CLINICAL TRIAL: NCT02304289
Title: Phase I Dose-Escalation Study Evaluating the Safety and Pharmacokinetics of Oral Artesunate (ART) in Patients With Advanced Hepatocellular Carcinoma (HCC).
Brief Title: Dose-Escalation Study Evaluating the Safety and Pharmacokinetics of Artesunate in Patients With Hepatocellular Carcinoma
Acronym: DESPARTH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow recruitment of patients
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO/2014/003; 2014-002503-16 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-12-01 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Artesunate (Experimental): The first patient will receive 200 mg Artesunate once-daily for 14 days. If no dose-limiting toxicity (DLT) is observed after 14 days, the next patient will start at a daily dose of 300 mg Artesunate. If no DLT is observed after 14 days, a cohort of 3 patients will receive 400 mg once-daily for 14 days. For each subsequent cohort of 3 patients 200 mg will be added to the dose, until the maximum tolerated dose (MTD) is determined.
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Oral Artesunate once-daily for 14 days, dose-escalation

SUMMARY:
The purpose of this study is to evaluate the Safety and Pharmacokinetics of Oral Artesunate in patients with advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Artemisinins, compounds extracted from the herb Artemisia annua, are safe and effective FDA-approved antimalarial drugs. Recent studies have suggested that artemisinins also exert anti-angiogenic and cytotoxic effects on human cancer cells. Artesunate (ART) is a water soluble semisynthetic artemisinin with improved pharmacokinetic properties.

A single-center phase I dose-escalation study evaluating the safety and pharmacokinetics of oral Artesunate in patients with Advanced HCC.

Approximately 15 patients will be enrolled in this trial. Dose-escalation protocol: The first patient will receive 200 mg Artesunate once-daily for 14 days. If no dose-limiting toxicity (DLT) is observed after 14 days, the next patient will start at a daily dose of 300 mg Artesunate. If no DLT is observed after 14 days, a cohort of 3 patients will receive 400 mg once-daily for 14 days. For each subsequent cohort of 3 patients 200 mg will be added to the dose, until the maximum tolerated dose (MTD) is determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced HCC, based on the report of the department of pathology, excluding fibrolamellar carcinoma.
* Liver mass measuring at least 2 cm with characteristic vascularization seen on either triphasic computed tomography (CT) scan or magnetic resonance imaging (MRI) with gadolinium
* Patients must have refused treatment with sorafenib or must have had treatment with sorafenib, which was either stopped due to intolerance or therapeutic failure.
* ECOG PS of 0-2.
* Child Pugh class ≤ B7
* Life expectancy greater than 3 months in the Investigator's opinion
* Adequate bone marrow function
* Adequate hepatic function
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin (β-hCG) or urine pregnancy test at screening. Women who are pregnant or breast feeding are ineligible for this study.
* For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use adequate methods of contraception (e.g., hormonal implants, combined oral contraceptives, vasectomized partner), during the treatment period and for at least 3 months after the last dose of study treatment
* For men: agreement to use a barrier method of contraception during the treatment period and for at least 3 months after the last dose of the study treatment.
* Adequate renal function
* Each subject (or their legally acceptable representative) must be able and willing to provide an written informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
* Able to swallow capsules
* Adequate coagulation tests: international normalized ratio (INR) ≤1.5 x ULN
* Recovery to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies
* At least 4 weeks since any major surgery or open biopsy and 7 days since a core biopsy before first study treatment
* The following time must have elapsed between previous therapy for cancer and first administration of ART:
* At least 2 weeks since previous systemic targeted therapy with small molecule inhibitors, which includes any tyrosine-kinase inhibitor
* At least 4 weeks since the last dose of systemic anti-cancer therapy other than targeted therapy, which includes cytotoxic agents, monoclonal antibody therapy, immunotherapy and prior radiotherapy

Exclusion Criteria:

* Patients with Child-Pugh classification > B7
* Major debilitating disease limiting survival prognosis (incl. heart failure, uncontrolled diabetes, psychiatric disease, hemodialysis, and respiratory insufficiency)
* Any mental deficiency preventing proper understanding of trial protocol requirements
* Remaining toxicities from previous sorafenib treatment will be individually evaluated and well documented by the PI.
* QTc≥440 msec
* Patients suffering from sinus bradycardia, bradyarrythmia, AV-block I or III.
* Known allergy to ART or to other artemisinin derivatives
* Malabsorption or intestinal obstruction
* History of venous thromboembolic disease within 3 months prior to first administration of study treatment
* The patient has current, severe and uncontrolled medical condition such as infection, diabetes mellitus or other systemic disease
* Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the drug
* The patient has known positive serology for human immunodeficiency virus
* Essential medications that are known potent inhibitors or inducers of CYP2B6 and/or CYP3A4
* Fibrolamellar carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 14 days
Maximum tolerated dose (MTD) | 14 days
Pharmacokinetic analysis of Cmax, Cmin, Tmax, and AUC. | 2 days

SECONDARY OUTCOMES:
Time to tumor progression (TTP) | Time from the first intake of Artesunate to radiological progression
Overall survival (OS) | ime from the first intake of Artesunate to death
Quality of life based on the "Functional Assessment of Cancer Therapy Hep-30 scale" (FACT-Hep-30) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Vlierberghe, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Dept. of Hepatology & Gastroenterology Ghent University Hospital, Ghent, East-Flandres, Belgium